CLINICAL TRIAL: NCT02747797
Title: Histology-Independent Study of the Multikinase Inhibitor Lucitanib (E3810) in Patients With Advanced Cancer and Fibroblast Growth Factor Receptor (FGFR), Vascular Endothelial Growth Factor Receptors (VEGFR), or Platelet Derived Growth Factor Receptor (PDGFR) Pathway Aberrations
Brief Title: Lucitanib (E3810) in Patients With Advanced Cancer and FGFR, VEGFR, or PDGFR Pathway Aberrations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug Supply No Longer Available
Sponsor: Teresa Helsten, MD (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Teresa Helsten, MD, Associate Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 141506
Record Dates: First submitted 2016-03-22; First posted 2016-04-22 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Lucitanib (E3810); Fibroblast Growth Factor Receptor; FGFR; Vascular Endothelial Growth Factor Receptor; VEGFR; Platelet Derived Growth Factor Receptor; PDGFR; metastatic malignancy
MeSH Terms: conditions — Acrocephalosyndactylia; Neoplasms | interventions — E-3810; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Advanced cancer with lucitanib-targeting biomarker(s) (Experimental): Lucitanib 10 mg orally daily
  Interventions: Drug: Lucitanib

INTERVENTIONS:
Drug: Lucitanib — 10 mg orally daily
  Other Names: E3810

SUMMARY:
Lucitanib is an oral multi kinase inhibitor designed to block the action of certain molecules called "angiogenic factors" that may cause tumors to grow. These factors are called vascular endothelial growth factor (VEGF), platelet derived growth factor receptor (PDGFR) and fibroblast growth factor (FGF). Lucitanib is experimental and not approved by the FDA for the treatment of cancer.

The purpose of this study is to look at the effects of lucitanib in cancer patients whose cancers harbor aberrations in FGFR, VEGFR, PDGFR or other markers predicted to be sensitive to lucitanib. This study will also look for biomarkers in samples of blood and tumor tissue to identify patients most likely to respond to lucitanib. Biomarkers are substances such as genetic material (DNA and RNA) and proteins found in blood and tumor tissue that might show if a cancer patient will respond or not respond to a drug.

DETAILED DESCRIPTION:
Lucitanib is an oral multi kinase inhibitor designed to block the action of certain molecules called "angiogenic factors" that may cause tumors to grow. These factors are called vascular endothelial growth factor (called VEGF), platelet derived growth factor receptor (PDGFR) and fibroblast growth factor (called FGF). Lucitanib is experimental and not approved by the FDA for the treatment of cancer.

The purpose of this clinical trial is to study the following in cancer patients whose cancers harbor aberrations in FGFR, VEGFR, PDGFR, or other biomarkers predicted to be sensitive to lucitanib:

* To look at the effects of lucitanib on their disease at 10 mg once daily.
* To look for biomarkers in samples of blood and tumor tissue to identify patients most likely to respond to lucitanib.
* To look at the safety of lucitanib in these patients

This is a two-center, open-label, non-randomized Phase II study of lucitanib in adult subjects with advanced cancers. Treatment will consist of daily oral administration of 10mg of lucitanib in 28-day cycles.

All patients providing informed consent will be screened for eligibility. Baseline assessments will include vital signs, physical exam, blood hematology and chemistries, ECG, and ECHO. If not done within the prior 4 weeks, a PET/CT scan, MRI, and/or CT scan will be performed for radiological evaluation of disease.

Clinical evaluations include physical exam, vitals, ECG (obtained once every month throughout treatment); blood hematology and chemistries (obtained every two weeks for the first three months and then once every month throughout treatment); radiologic evaluations (PET/CT, CT and/or MRI, +/- bone imaging as clinically appropriate) will be performed every 8 weeks.

This study may last up to approximately 4 years or longer, depending on whether or not the study doctor feels that continuing lucitanib dosing is in the patient's best interest. Once a patient finishes study treatment with lucitanib, patients will need to complete an End of Study visit. Each of the study visits can last from approximately 2 to 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed advanced or metastatic malignancy characterized by one or more of the following:

  * Subject is intolerant of standard therapy
  * Malignancy is refractory to standard therapy
  * Malignancy relapsed after standard therapy
  * Malignancy for which there is no standard therapy that improves survival by at least 3 months.
* Subjects must have evaluable tumor(s) with documented alteration(s) in potential lucitanib related biomarker(s) VEGFR, FGFR, PDGFR.
* Laboratory function within specified parameters:

  * Adequate bone marrow function: absolute neutrophil count ≥ 1,500/mL; hemoglobin ≥ 8.5 g/dL, platelets ≥ 75,000/mL.
  * Adequate liver function: transaminases (AST/ALT) and alkaline phosphatase ≤ 3 (≤ 5 X ULN in the setting of liver metastasis) x ULN; bilirubin ≤ 1.5 x ULN.
  * Adequate renal function: creatinine clearance ≥ 40 mL/min (Cockcroft Gault).
  * Adequate blood coagulation: international normalized ratio (INR) ≤ 2.3.
  * Serum amylase and lipase ≤ 1.5 x ULN.
* Adequately controlled blood pressure (BP): BP ≤ 150/90 mm Hg. Use of > 2 antihypertensive agents at enrollment is not allowed.
* Adequate performance status: Eastern Cooperative Oncology Group (ECOG) 0-2
* Subjects must be off other anti-tumor agents for at least 5 half lives of the agent or 4 weeks from the last day of treatment, whichever is shorter. Endocrine therapies (e.g., for breast or prostate cancer) and anti-Her2 therapies (for example, trastuzumab, pertuzumab, or lapatinib) are allowed to continue while on this study. Bisphosphonates or denosumab are allowed for subjects with bone metastasis.
* Subjects may not be receiving any other experimental agents or agents that are not FDA approved.

Exclusion Criteria:

* Pregnant or lactating women.
* Uncontrolled hypertension (defined as SBP ≥ 140 mmHg and/or DBP ≥ 90 mmHg with optimized antihypertensive therapy)
* Subjects who have not recovered from toxicities as a result of prior anticancer therapy, except alopecia and infertility. Recovery is defined as < Grade 2 severity per Common Terminology Criteria for Adverse Events Version 4.3.
* Significant cardiovascular impairment: history of CHF greater than New York Heart Association (NYHA) Class II, unstable angina, MI or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment.
* Uncontrolled hypothyroidism defined as serum TSH higher than 5 mIU/mL while receiving appropriate thyroid hormone therapy.
* Bleeding or thrombotic disorders or use of anticoagulants requiring therapeutic INR monitoring, e.g., warfarin or similar agents. Treatment with LMWH and factor X inhibitors that do not require INR monitoring is permitted. Anti-platelet agents are prohibited throughout the study.
* Current treatment with any prohibited medications associated with prolongation of QT interval.
* Received strong inhibitors of CYP2C8 or CYP3A4 or strong inducers of CYP3A4 ≤ 7 days prior to first dose of lucitanib or have on-going requirements for these medications.
* Received bevacizumab < 3 months prior to first dose of lucitanib.
* Major surgery (not including placement of central lines) within 3 weeks prior to study or planned surgery during the course of this study.
* Subjects with breast or lung cancer who are eligible for other clinical trials of lucitanib open at their institution are not eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Response rates to lucitanib in subjects with advanced cancers harboring aberrations targeted by lucitanib. | 28-day cycle

SECONDARY OUTCOMES:
Clinical Benefit rates (complete response (CR), partial response (PR), or stable disease (SD) ≥ 6 months) in the study population. | through study completion, up tp 3 years
  Clinical Benefit will be defined as SD ≥ 6 cycles and PR/CR of any duration.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28-day cycle
  Toxicities will be described according to the NCI-CTCAE Version 4.3. Unacceptable toxicity is defined as any clinically significant Grade 3 or 4 toxicity including expected toxicities definitely, probably, or possibly related to the study medication that are not amenable to dose reduction
Correlation between response rates and specific molecular tumor profile (type of FGF/FGFR or other aberration) in a descriptive fashion | 28-day cycle

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Helsten, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States